CLINICAL TRIAL: NCT03820440
Title: End-expiratory Occlusion Test and Lung Recruitment Maneuver to Assess Fluid responsiVeness In Surgical Patients: an Open-label, Randomized Clinical Trial
Brief Title: End-expiratory Occlusion Test and Lung Recruitment Maneuver to Assess Fluid responsiVeness In Surgical Patients
Acronym: ELVIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Antonio Messina, ICU senior consultant, Humanitas Clinical and Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ELVIS
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hemodynamic Instability; Surgery; Fluid Overload
Keywords: End-expiratory occlusion test; Lung Recruitment Manovre; Fluid responsiveness; Functional Hemodynamic Test
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: The study protocol is started during a period of intraoperative hemodynamic stability, as previously defined (change in mean arterial pressure of less than 10% during 5 minutes). The study protocol is the following: 1) a set of measurements is recorded (T0) at a baseline ventilation of 7 ml/Kg and then the EEOT is performed by using the software function, "expiratory hold", to interrupt mechanical ventilation; 2) after one minute a set of measurements was recorded (T1); 3) the LRM is then performed; 4) after one minute another set of measurements is recorded (T2) and then a fluid challenge of 4 mL/Kg of crystalloid solution is infused over 10 minutes. The attending anesthetist is allowed to interrupt the protocol at any stage for either hemodynamic instability or any other adverse effects requiring urgent treatment. The sequence of application of EEOT and LRM on the same patient (EEOT_LRM or LRM_EEOT) is randomly generated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment - hemodynamic tests (Experimental): Treatment - hemodynamic tests:
  The EEOT is performed by interrupting the mechanical ventilation for 30 seconds, by using and end-expiratory hold on the ventilator.
  The LRM is performed by using a single act of mechanical ventilation in pressure-controlled mode at 30 cmH20 for 30 seconds
  Interventions: Diagnostic Test: End-expiratory occlusion test (EEOT); Diagnostic Test: Lung recruitment manovre (LRM)

INTERVENTIONS:
Diagnostic Test: End-expiratory occlusion test (EEOT) — The EEOT is performed by interrupting the mechanical ventilation for 30 seconds, by using and end-expiratory hold on the ventilator.
Diagnostic Test: Lung recruitment manovre (LRM) — The LRM is performed by using a single act of mechanical ventilation in pressure-controlled mode at 30 cmH20 for 30 seconds

SUMMARY:
The functional hemodynamic test (FHT) called passive leg raising (PLR) has been successfully used for assessing the fluid responsiveness in ICU patients since 2009 and its reliability has been confirmed by three large meta-analyses. However, the PLR is not usually practicable in the OR.

A lot of different FHTs have been proposed, as alternative to the PLR, in ICU and, more recently, OR. These tests could be basically subdivided in two groups. A subgroup of FHTs is based on sudden and brief variations of the mechanical ventilation to induce a change in right ventricle preload and/or after load and, as consequence, of left ventricle SV. A second subgroup aims at testing the increase in SV after the rapid administration of a small aliquot of the predefined FC.

Among the first group, the end-expiratory occlusion test (EEOT) and the lung recruitment maneuver (LRM) have been previously successfully tested in surgical patients. The EEOT consists of the interruption of the mechanical ventilation for 30 seconds, whereas the LRM consists in the increase in the peak inspiratory pressure up to 30 cmH20 for 30 seconds and in the assessment of the changes in the SV after the maneuvers. These tests are safe and can be easily applicable during the surgery to predict fluid responsiveness and optimize the fluid therapy.

The primary aim of the present study is to compare the reliability of EEOT and LRM in predicting fluid responsiveness in patients undergoing general surgery.

DETAILED DESCRIPTION:
Targeted fluid therapy has received increasing attention in the management of patients showing acute circulatory failure in both intensive care unit (ICU) and operating room (OR), aiming at preventing both inadequate tissue blood flow and fluid overload [1]. In fact, unnecessary fluid administration can increase morbidity and mortality and length of hospital stay of critically ill and surgical patients [2-10].

Since the only physiological reason to give a fluid challenge (FC) is to increase the stroke volume (SV) [11-13] and this effect is obtained only in about 50% of ICU and OR patients [14, 15], a vast literature investigated the possibility of predict this effect before FC administration, but the issue remains extremely challenging [1, 13, 16-18]. Bedside clinical signs and pressure and static volumetric static variables, do not predict fluid responsiveness [17]. Moreover, several physiological factors affect the reliability of the ventilator-induced dynamic changes in pulse pressure and stroke volume [pulse pressure variation (PPV) and stroke volume variation (SVV), respectively], and their echographic surrogates, in a significant number of ICU and OR patients [19-22].

To overcome these limitations, the functional hemodynamic assessment (i.e. the assessment of the dynamic interactions of hemodynamic variables in response to a defined perturbation), of fluid responsiveness has gained in popularity [17, 18, 23]. A functional hemodynamic test (FHT) consist in a manoeuvre determining a sudden change in cardiac function and/or heart lung interaction, affecting the hemodynamics of fluid responders and non-responders to a different extent [17, 18, 23].

The FHT called passive leg raising (PLR) has been successfully used for assessing the fluid responsiveness in ICU patients since 2009 [24] and its reliability has been confirmed by three large meta-analyses [25-27]. However, the PLR is not usually practicable in the OR.

A lot of different FHTs have been proposed, as alternative to the PLR, in ICU and, more recently, OR. These tests could be basically subdivided in two groups. A subgroup of FHTs is based on sudden and brief variations of the mechanical ventilation to induce a change in right ventricle preload and/or after load and, as consequence, of left ventricle SV [24, 28]. A second subgroup aims at testing the increase in SV after the rapid administration of a small aliquot of the predefined FC [29, 30].

Among the first group, the end-expiratory occlusion test (EEOT) and the lung recruitment maneuver (LRM) have been previously successfully tested in surgical patients [31-33]. The EEOT consists of the interruption of the mechanical ventilation for 30 seconds, whereas the LRM consists in the increase in the peak inspiratory pressure up to 30 cmH20 for 30 seconds and in the assessment of the changes in the SV after the maneuvers. These tests are safe and can be easily applicable during the surgery to predict fluid responsiveness and optimize the fluid therapy.

The primary aim of the present study is to compare the reliability of EEOT and LRM in predicting fluid responsiveness in patients undergoing general surgery.

(for Bibliography please refer to the original protocol)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥ 18 years;
2. Scheduled for elective supine abdominal surgery and requiring invasive arterial monitoring;
3. Glasgow coma scale 15 at recruitment. All the patients must be able to sign an informed consent at the admission.

Exclusion Criteria:

1. Any recurrent cardiac arrhythmias;
2. Reduced left (ejection fraction <30%) or right (systolic peak velocity of tricuspid annular motion <0.17 m/s) ventricular systolic function;
3. Chronic use beta-blocking agents.
4. History of pneumothorax.
5. BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC difference | 10 minutes after fluid challenge administration
  To assess the difference in the area under (AUC) the receiving operator characteristic curve (ROC)

SECONDARY OUTCOMES:
Sensitivity and Specificity | 10 minutes after fluid challenge administration
  ROC curve analysis to assess the sensitivity and specificity of EEOT and LRM in predicting fluid responsiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Biais M, Larghi M, Henriot J, de Courson H, Sesay M, Nouette-Gaulain K. End-Expiratory Occlusion Test Predicts Fluid Responsiveness in Patients With Protective Ventilation in the Operating Room. Anesth Analg. 2017 Dec;125(6):1889-1895. doi: 10.1213/ANE.0000000000002322. PMID 28742783
- [Result] Biais M, Lanchon R, Sesay M, Le Gall L, Pereira B, Futier E, Nouette-Gaulain K. Changes in Stroke Volume Induced by Lung Recruitment Maneuver Predict Fluid Responsiveness in Mechanically Ventilated Patients in the Operating Room. Anesthesiology. 2017 Feb;126(2):260-267. doi: 10.1097/ALN.0000000000001459. PMID 27922547